CLINICAL TRIAL: NCT04985864
Title: A Study on Effect of Simultaneous Application of Transcranial Direct Current Stimulation (tDCS) and Robotic Gait Training on Gait Function in Stroke Patients With Gait Impairment
Brief Title: Effect of Simultaneous Application of HD-tDCS and Robot-assisted Gait Training on Gait Function in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yun-Hee Kim (Other)
Collaborators: Ybrain Inc. (Industry)
Responsible Party: Sponsor-Investigator, Yun-Hee Kim, Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-06-131
Record Dates: First submitted 2021-07-19; First posted 2021-08-02 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot gait training with brain stimulation (Experimental): Lokomat robot training and anodal transcranial direct current stimulation (tDCS) on the leg motor areas
  Interventions: Device: Brain stimulation; Device: Treadmill gait training
- Gait training with sham brain stimulation (Active Comparator): Treadmill gait training and anodal sham transcranial direct current stimulation (tDCS) on the leg motor areas
  Interventions: Device: Treadmill gait training

INTERVENTIONS:
Device: Brain stimulation — tDCS brain stimulation on leg motor areas was applied to stroke patients.
  Arms: Robot gait training with brain stimulation
Device: Treadmill gait training — Lokomat robot training was applied to stroke patients.

SUMMARY:
The purpose of this study was to investigate the effects of simultaneous application of transcranial direct current stimulation (tDCS) with robotic gait training in stroke patients with gait impairment.

ELIGIBILITY:
Inclusion Criteria:

* Age: 19 - 79 years
* More than 3 months post stroke
* Functional ambulation classification (FAC) (1~4)

Exclusion Criteria:

* History of serious neurological disease other than stroke
* Difficult to understand experimental tasks because of extremely severe cognitive impairment (Korean-Mini-Mental State Examination, K-MMSE≤10)
* History of psychiatric disease
* Contraindicated to tDCS

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Change in 10 meter walk test | session 0 (initial visit); session 10 (at approximately 4 weeks); after 4 weeks from intervention termination (follow-up)
  Measurement of the time it takes a subject to walk 10m with self selected gait speed. To perform the test, patient walks 10 meters (33 ft) and the time is measured when the leading foot crosses the start line and the finish line. The instructions are: "Please walk this distance at your normal pace when I say go."

SECONDARY OUTCOMES:
Change in Berg Balance Scale (BBS) | session 0 (initial visit); session 10 (at approximately 4 weeks); after 4 weeks from intervention termination (follow-up)
  Measurement of balance function. A five-point ordinal scale, ranging from 0-4. "0" indicates the lowest level of function and "4" the highest level of function. Score the lowest performance. Total Score = 56.
Change in Timed Up and Go test (TUG) | session 0 (initial visit); session 10 (at approximately 4 weeks); after 4 weeks from intervention termination (follow-up)
  11-20 seconds are within normal limits for frail elderly and disabled patients, and greater than 20 seconds means the person needs assistance outside and indicates further examination and intervention. A score of 30 seconds or more suggests that the person may be prone to falls.
Changes in Brain activation of resting-state functional MRI | session 0 (initial visit); session 10 (at approximately 4 weeks)
  Measure of Neuroplasticity
Change in Geriatric Depression Scale (GDS) | session 0 (initial visit); session 10 (at approximately 4 weeks); after 4 weeks from intervention termination (follow-up)
  Measure of depression. The grid sets a range of 0-9 as "normal", 10-19 as "mildly depressed", and 20-30 as "severely depressed".
Changes in motor evoked potential | session 0 (initial visit); session 10 (at approximately 4 weeks); after 4 weeks from intervention termination (follow-up)
  Resting motor threshold (rMT) and amplitude of motor evoked potential in first dorsal interosseous muscle are measured. These outcomes are measured by transcranial magnetic stimulation over the motor hotspot. The rMT is defined as the minimum stimulus intensity that produced a minimal motor evoked response at rest. The amplitude means peak to peak of the muscle response.
Change in Fugl-Meyer Assessment | session 0 (initial visit); session 10 (at approximately 4 weeks); after 4 weeks from intervention termination (follow-up)
  The score is a stroke-specific, performance-based impairment index. The degree of impairment of upper and lower limbs is measured.
Change in Functional ambulatory category | session 0 (initial visit); session 10 (at approximately 4 weeks); after 4 weeks from intervention termination (follow-up)
  The Functional Ambulation Categories (FAC) is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device. The higher the score, the better the walking ability.
Change in Modified Bathel index (MBI) | session 0 (initial visit); session 10 (at approximately 4 weeks); after 4 weeks from intervention termination (follow-up)
  The MBI is a measure of activities of daily living, which shows the degree of independence of a patient from any assistance. It covers 10 domains of functioning (activities): bowel control, bladder control, as well as help with grooming, toilet use, feeding, transfers, walking, dressing, climbing stairs, and bathing.
Change in Muscle Manual Test (MMT) | session 0 (initial visit); session 10 (at approximately 4 weeks); after 4 weeks from intervention termination (follow-up)
  Manual muscle testing (MMT) is a procedure for the evaluation of the function and strength of individual muscles and muscle groups based on the effective performance of a movement in relation to the forces of gravity and manual resistance.
Change in Range of Motion (ROM) | session 0 (initial visit); session 10 (at approximately 4 weeks); after 4 weeks from intervention termination (follow-up)
  Range of Motion (ROM) testing is the measurement of movement around a specific joint or body part.
Change in Modified Ashworth Scale(MAS) | session 0 (initial visit); session 10 (at approximately 4 weeks); after 4 weeks from intervention termination (follow-up)
  measures spasticity with scale from 0 to 3. 0 is no increase in muscle tone. 3 is considerable increase in muscle tone, passive movement difficult.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea